CLINICAL TRIAL: NCT02625545
Title: Study of Median Lobe Prostatic UroLift Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeoTract, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP00001
Record Dates: First submitted 2015-12-05; First posted 2015-12-09 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UroLift System procedure (Experimental): All eligible,enrolled subjects will undergo a UroLift procedure
  Interventions: Device: UroLift System procedure

INTERVENTIONS:
Device: UroLift System procedure — Minimally invasive procedure for treatment of lower urinary tract symptoms (LUTS) due to BPH
  Other Names: Prostatic UroLift (PUL)

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of using UroLift in subjects with a prostatic median lobe enlargement due to benign prostatic hyperplasia (BPH).

DETAILED DESCRIPTION:
Study Objectives: Evaluate the safety and effectiveness of the UroLift® System when used in symptomatic benign prostatic hyperplasia (BPH) subjects with an enlarged median lobe.

Study Design: Prospective, multicenter, non-blinded, single arm (non-randomized) study.

Sample Size: A total of no more than 48 subjects will be enrolled. Subject Population: Males age of 50 years or older diagnosed with lower urinary tract symptoms (LUTS) with enlarged median lobe.

ELIGIBILITY:
Inclusion Criteria:

* Enlarged median lobe (ML) contributing to obstruction of the prostate
* BPH

Exclusion Criteria:

-

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-02-17 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan B. Rukstalis, M.D., Principal Investigator — Wake Forest

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | UroLift System Procedure
Started | 45
3 Month | 45
6 Month | 45
12 Month | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat (analysis population)
Groups:
- UroLift Arm: Subjects that undergo the UroLift System procedure.
Arm/Group | UroLift Arm
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 40
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 45
IPSS Baseline [Mean (Standard Deviation); unit: Scores on a scale] — The International Prostate Symptom Score (IPSS) is a standardized 8 question (7 symptom questions + 1 quality of life question) written screening tool used to screen for, rapidly diagnose, track the symptoms of, and suggest management of the symptoms of the disease benign prostatic hyperplasia (BPH). The symptoms must have been experienced in the last month and each answer is scored from 0 to 5 for a maximum score of 35 points.Those patients scoring 7 or below are generally considered mildly symptomatic, whereas 20 or above is considered severely symptomatic.
  Scores on a scale | 24.2 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: At 6 Months, the 95% Lower Confidence Limit of the Mean Percent Improvement in IPSS Over Baseline for the UroLift System Must be ≥ 25%.
Description: The International Prostate Symptom Score (IPSS) is a standardized 8 question (7 symptom questions + 1 quality of life question) written screening tool used to screen for, rapidly diagnose, track the symptoms of, and suggest management of the symptoms of the disease benign prostatic hyperplasia (BPH). The symptoms must have been experienced in the last month and each answer is scored from 0 to 5 for a maximum score of 35 points.Those patients scoring 7 or below are generally considered mildly symptomatic, whereas 20 or above is considered severely symptomatic.
Time Frame: 6 months
Population: Intent to treat Population
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | UroLift System Procedure
Number analyzed (Participants) | 45
percent change | 57.7 [50.8 to 63.8]

2. Secondary Outcome: Intent to Treat Population International Prostate Symptom Scores at Baseline and 12 Month Follow-up
Description: as for outcome 1
Time Frame: 12 Months
Population: 44/45, 1 Subject was retreated with additional UroLift System devices prior to the 12 month Follow up visit.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | UroLift System Procedure
Number analyzed (Participants) | 44
Score on a scale
  Baseline IPSS | 24.1 (5.0)
  12 Month IPSS | 10.6 (7)

3. Secondary Outcome: Intent to Treat Population International Prostate Symptom Score Percent Change From Baseline to 12 Month Follow-up
Description: Present change in Intent to Treat population International Prostate Symptom Score (IPSS) from Baseline to 12 Month Follow-up
Time Frame: 12 Months
Population: 44/45, 1 Subject was retreated with additional UroLift System devices prior to the 12 month Follow-up visit.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | UroLift System Procedure
Number analyzed (Participants) | 44
percent change | -55.1 [-63.6 to -46.6]

4. Secondary Outcome: Intent to Treat Population Quality of Life Scores at Baseline and 12 Month Follow-up
Description: Quality of Life (QOL) score results from a disease-specific (BPH) quality of life question (bother score) scored on a scale from 0 to 6 points (delighted to terrible).
Time Frame: 12 Months
Population: 44/45, 1 Subject was retreated with additional UroLift System devices prior to the 12 month Follow-up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | UroLift System Procedure
Number analyzed (Participants) | 44
score on a scale
  Baseline QOL | 4.9 (0.8)
  12 Month QOL | 1.9 (1.3)

5. Secondary Outcome: Intent to Treat Population Quality of Life Score Perfect Change From Baseline to 12 Month Follow-up
Description: as for outcome 4
Time Frame: 12 Months
Population: 44/45, 1 Subject was retreated with additional UroLift System devices prior to the 12 month Follow-up visit.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | UroLift System Procedure
Number analyzed (Participants) | 44
percent change | -61.1 [-69.5 to -52.7]

6. Secondary Outcome: Intent to Treat Population BPHII Scores at Baseline and 12 Month Follow-up
Description: BPHII (Benign Prostatic Hyperplasia Impact Index) is used to assess the impact of BPH symptoms on subject health and functioning. The BPHII is a self-administered questionnaire with 4 questions about urinary problems during the past month regarding physical discomfort, worry about health, how bothersome symptoms are, and whether the symptoms are interfering with doing usual activities. Scores for each question range from 0 to 4, with higher score indicating greater impact. Maximum score is 16.
Time Frame: 12 Months
Population: 44/45, 1 Subject was retreated with additional UroLift System devices prior to the 12 month Follow-up visit.
Measure: Mean (Standard Deviation); unit: BPHII score
Arm/Group | UroLift System Procedure
Number analyzed (Participants) | 44
BPHII score
  Baseline BPHII | 7.7 (2.8)
  12 Month BPHII | 2.1 (2.5)

7. Secondary Outcome: Intent to Treat Population BPHII Score Percent Change From Baseline to 12 Month Follow-up
Description: Present change in Intent to Treat population, Benign Prostatic Hyperplasia Impact Index (BPHII) score from Baseline to 12 Month Follow-up
Time Frame: 12 Months
Population: 44/45, 1 Subject was retreated with additional UroLift System devices prior to the 12 month Follow-up visit.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | UroLift System Procedure
Number analyzed (Participants) | 44
percent change | -70.4 [-81.9 to -59.0]

8. Secondary Outcome: Intent to Treat Population Peak Flow Rate Scores at Baseline and 12 Month Follow-up
Description: Peak or maximum flow rate [ml/sec] was collected using uroflowmetry, a standard diagnostic used to test to assess how well the urinary tract functions. A lower number indicates a reduced flow rate.
Time Frame: 12 Months
Population: 37/45, 1 Subject was retreated with additional UroLift System devices prior to the 12 month Follow-up visit. Includes only cases where voided volume is at least 125ml.
Measure: Mean (Standard Deviation); unit: mL/sec
Arm/Group | UroLift System Procedure
Number analyzed (Participants) | 37
mL/sec
  Baseline Qmax | 7.1 (2.7)
  12 Month Qmax | 13.5 (7.6)

9. Secondary Outcome: Intent to Treat Population Peak Flow Rate Percent Change From Baseline to 12 Month Follow-up
Description: as for outcome 8
Time Frame: 12 Months
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | UroLift System Procedure
Number analyzed (Participants) | 37
percent change | 108.4 [64.0 to 152.8]

10. Secondary Outcome: Intent to Treat Population Post Void Residual Measurement at Baseline and 12 Month Follow-up
Description: Post Residual Void (PVR) is the amount of urine left in the bladder after using the restroom. PVR is determined using ultrasound or bladder scanner.
Time Frame: 12 Months
Population: 44/45, 1 Subject was retreated with additional UroLift System devices prior to the 12 month Follow-up visit.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | UroLift System Procedure
Number analyzed (Participants) | 44
mL
  Baseline PVR | 108.5 (80.5)
  12 Month PVR | 69.9 (77.0)

11. Secondary Outcome: Intent to Treat Population Post Void Residual Change From Baseline to 12 Month Follow-up
Description: as for outcome 10
Time Frame: 12 Months
Population: 44/45, 1 Subject was retreated with additional UroLift System devices prior to the 12 month Follow-up visit.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | UroLift System Procedure
Number analyzed (Participants) | 44
percent change | -4.8 [-38.1 to 28.4]

ADVERSE EVENTS:
Time Frame: 12 Months
Description: Adverse Events reported from Index Procedure through 12 Months follow-up; No Unexpected Adverse Device Events
Arm/Group | UroLift System Procedure
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 5/45
Other Adverse Events (participants affected / at risk) | 36/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UroLift System Procedure (N=45)
Bradycardia/Heartblock (Cardiac disorders) | 1 (1)
Cervical spinal stenosis (Nervous system disorders) | 1 (1) — cervical spinal stenosis cord compression
Pain in hip (Musculoskeletal and connective tissue disorders) | 1 (1) — Right Hip Pain
Urinary tract infection (Gastrointestinal disorders) | 1 (1)
Aspiration pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UroLift System Procedure (N=45)
Haemorrhage urinary tract (Renal and urinary disorders) | 26 (27) — blood clot in urine
Dysuria (Renal and urinary disorders) | 22 (22)
Hematuria (Renal and urinary disorders) | 12 (13)
Micturition urgency (Renal and urinary disorders) | 4 (4) — Urinary urgency
Urinary tract infection (Infections and infestations) | 7 (8)
Ejaculation disorder (Reproductive system and breast disorders) | 3 (3)
Urge incontinence (Renal and urinary disorders) | 3 (3)
Urinary retention (Renal and urinary disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT02625545/Prot_SAP_001.pdf